CLINICAL TRIAL: NCT05820139
Title: A Randomized Controlled Single-Blinded Study Evaluating the Optimal Volume Voided for Passage of a Backfill-Assisted Voiding Trial Following Urogynecologic Surgery
Brief Title: Evaluating the Optimal Volume Voided for Passage of a Backfill-Assisted Voiding Trial Following Urogynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00091698
Record Dates: First submitted 2023-04-07; First posted 2023-04-19 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Voiding Dysfunction
Keywords: Urinary Tract Infections; overactive bladder; pelvic organ prolapse surgery; urinary incontinence surgery
MeSH Terms: conditions — Urinary Tract Infections; Urinary Bladder, Overactive | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be recruited at an Urogynecology office either at the pre-operative visit or on the day of surgery
Who Masked: Participant
Masking Description: The voiding trial instructions for each specific patient will be given to the Post Anesthesia Care Unit (P(ACU) or floor Registered Nurse (RN) taking care of the patient and will include what volume voided equals a passing voiding trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (voids 2/3 of the volume backfilled) (Other): control group
  Interventions: Procedure: Control Group
- test group (voids ½ of the total volume backfilled) (Active Comparator): test group)
  Interventions: Procedure: Test Group

INTERVENTIONS:
Procedure: Control Group — Patients will be randomized to a 200mL (control group)
  Other Names: backfill-assisted voiding trial
  Arms: control group (voids 2/3 of the volume backfilled)
Procedure: Test Group — Patients will be randomized to a cut-off of 150mL (test group)
  Other Names: backfill-assisted voiding trial
  Arms: test group (voids ½ of the total volume backfilled)

SUMMARY:
Urinary retention can lead to bladder over-distention, ischemia, and long-term voiding dysfunction, and early identification of urinary retention can help prevent these adverse events

DETAILED DESCRIPTION:
Postoperative voiding trials (VT) can identify as well as prevent postoperative urinary retention. Voiding trial protocols vary by provider and healthcare facilities/institutions as there is no consensus on how to prevent postoperative urinary retention optimally. Identification of an optimal VT could not only help decrease adverse events associated with urinary retention but also decrease postoperative catheter-associated urinary tract infection (CAUTI) rates, unplanned hospital or clinic visits, and decrease patient discomfort while increasing patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant women >18yo undergoing pelvic organ prolapse or urinary incontinence surgery

Exclusion Criteria:

* Patients undergoing fistula repair or sacral neuromodulation
* Voiding dysfunction preoperatively that requires intermittent self-catheterization
* Intraoperative bladder injury
* Pregnancy
* Preoperative UTI (culture proven within 7 days prior to surgery)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pelvic organ prolapse or urinary incontinence
Enrollment: 100 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
difference in acute voiding dysfunction between a backfill assisted voiding trial | Week 6
  difference in acute voiding dysfunction between a backfill assisted voiding trial with a volume voided cutoff of 150mL vs. 200mL for passage of VT - Acute voiding dysfunction is defined as a failed voiding trial requiring discharge home with a catheter, as well as voiding dysfunction occurring at a later time that results in an emergency department/urgent care/clinic visit requiring either an indwelling catheter or clean intermittent catheterization (CIC)

SECONDARY OUTCOMES:
proportion of patients develops postoperative UTIs | Day 7
  UTI diagnosed by symptomatology alone or urinalysis (UA) + culture proven within one week (7 days) of catheter removal
proportion of patients developing overactive bladder symptoms | Week 6
  Sudden urge to urinate that is difficult to hold, with leakage of urine (even if you just voided recently), Frequent urination (>8 times/day), or waking up at night to urinate (2 or more times/night)
proportion of patients developing bladder pain or pressure | Week 6
  Bladder pain (pain or discomfort in the lower abdomen when your bladder is full) or bladder pressure (continuous feeling of pressure, not relieved by urination)
proportion of patients requiring repeat outpatient voiding trials | Week 6
  proportion of patients requiring repeat outpatient voiding trials
average number of days postoperatively, that require catheterization | Week 6
  average number of days postoperatively, that require catheterization

CONTACTS AND LOCATIONS:
Overall Officials: David Lovejoy, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT05820139/ICF_000.pdf